CLINICAL TRIAL: NCT02408809
Title: The Impact of Orthopaedic Smoking Cessation Education on Cigarette Abstinence Self-Efficacy: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Nkemakolam Egekeze, Orthopaedic Surgery Researcher, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15-247
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Cigarette Smoking
Keywords: Orthopaedic Smoking Cessation Discussion; Smoking Cessation; Randomized Controlled Trial
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator)
  Interventions: Behavioral: General Smoking Cessation Discussion
- Intervention (Active Comparator)
  Interventions: Behavioral: Orthopaedic Related Smoking Cessation Discussion

INTERVENTIONS:
Behavioral: General Smoking Cessation Discussion — This group receives the 5 A's of smoking cessation counseling incorporating how cigarette smoking negatively impacts general health (cancer, MI). 10 minutes in length.
  Arms: Control
Behavioral: Orthopaedic Related Smoking Cessation Discussion — The participants in this group receive a discussion including the 5 A's of smoking cessation counseling incorporating an orthopaedic related smoking cessation discussion about the effects of smoking cigarettes on the musculoskeletal system. 10 minutes in length.
  Arms: Intervention

SUMMARY:
The investigators of this study aim to evaluate the impact of a new orthopaedic related smoking cessation discussion on smoking behavior. Considering the high prevalence of patients who smoke and receive orthopaedic management, we are interested in determining whether an orthopaedic smoking cessation discussion impacts smoking abstinence self-efficacy over time compared to a general smoking cessation discussion.

ELIGIBILITY:
Inclusion Criteria:

* Daily cigarette smokers (5 cigarettes or more a day for past year), 18 years of age or older, new orthopaedic management, native English speaker

Exclusion Criteria:

* Patients unable to provide consent, suffer an impairment (mental, psychiatric, hearing or sight), alcohol and illicit drug abusers, homeless, presently managed with a smoking cessation medication or counseling, living with a cigarette smoker, user of other tobacco products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
SASEQ | 5 minutes
  Smoking abstinence Self-Efficacy Questionnaire

SECONDARY OUTCOMES:
Patient Knowledge and Motivation to Quit | less than 20 minutes
  Knowledge and Motivation assessments

CONTACTS AND LOCATIONS:
Overall Officials: Nkem Egekeze, MD, Principal Investigator — UMKC DEPT OF ORTHOPAEDIC SURGERY; Akin Cil, MD, Study Director — UMKC DEPT OF ORTHOPAEDIC SURGERY; Karen Williams, PhD, Study Director — UMKC DEPT OF BIOINFORMATICS; James Bogener, MD, Study Director — UMKC DEPT OF ORTHOPAEDIC SURGERY; Mark Bernhardt, MD, Study Director — UMKC DEPT OF ORTHOPAEDIC SURGERY; Jonathan Dubin, MD, Study Director — UMKC DEPT OF ORTHOPAEDIC SURGERY